CLINICAL TRIAL: NCT03209336
Title: Single Center Study of Intraoperative Radiotherapy for Middle and Low Rectal Cancer in the Standard of Peritoneal Inversion Rectal Cancer.
Brief Title: Study of Intraoperative Radiotherapy for Middle and Low Rectal Cancer
Acronym: IROT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Hospital of Jilin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SecondJilinU-IORT
Record Dates: First submitted 2017-06-30; First posted 2017-07-06 (Actual); Last update posted 2017-07-06 (Actual); Status verified 2017-07

CONDITIONS: Rectal Cancer
Keywords: Ultra-low rectal cancer; Intersphincteric resection; IORT
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A group (Experimental): Colorectal cancer patients first are given antineoplastic drugs and then transfer to operative room to be treated by surgical resection and the radiotherapy is given during the operation after the removal of the tumour.
  Interventions: Radiation: Intraoperative radiotherapy by Intrabeam（Zeiss Meditech，Jena，Germany）
- B group (No Intervention): Colorectal cancer patients first are given antineoplastic drugs and then transfer to operative room to be treated only by surgical resection and no radiotherapy afer the removal of the tumour.

INTERVENTIONS:
Radiation: Intraoperative radiotherapy by Intrabeam（Zeiss Meditech，Jena，Germany） — We confirmed that if the patients had the distant metastasis before IORT. The median radiation dose was 5.00 Gy (range: 5.00-10.00Gy), the average dose was 6.00 Gy. The median radiation time was 0:33:24 (range: 0:21:45-1:06:23), which was the same with the patients'. All patients' surface dose ranged from 15.00 to 28.50 Gy.
  Arms: A group

SUMMARY:
To study the application of Intersphincteric Resection（ISR）combined with intraoperative radiation therapy(IORT) for ultra-low rectal cancer,and to broaden the surgical indications of Intersphincteric Resection（ISR.

The study is aimed to assess the postoperative acute complication and the short-term acute efficacy on the patients with middle and low rectal cancer by treated with intraoperative radiotherapy,especially those with peritoneal inversion rectal cancer.

DETAILED DESCRIPTION:
Abstract objective: To study the application of Intersphincteric Resection（ISR）combined with intraoperative radiation therapy(IORT) for ultra-low rectal cancer,and to broaden the surgical indications of Intersphincteric Resection（ISR）.

Methods: Patients, who were diagnosed with ultra-low rectal cancer and had strong desire of preserving anal function, will take part in the research,whose tumor invading the levator ani muscle or above, the diameter less than 6cm, the lower tumor margin away from the anal verge by less than 5cm and away from the dentate line by less than 3cm.They will undergo total mesorectal excision(TME) and ISR combined with IORT and prophylactic ileostomy.

Outcomes Measures:The evaluation of short term effects includes complications such as anastomotic leakage, acute radiation injury ,urinary dysfunction ,dysfunction of anal sphincter ,sexual dysfunction ,local recurrence , total life expectancy and expectancy without metastasis. The postoperative pathological examination reported to be moderately differentiated adenocarcinoma .We wili assess their postoperative acute complications and short-term efficacy .Their time of follow up visit wil be 1 year or more.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria:

* Aged 40 to 80 years old, gender not limited.
* Be diagnosed as colorectal cancer by coloscopy.
* Patients with middle and low rectal cancer,whose preoperative staging evaluation is T3 ,T4 or N+.
* Accept surgery and intraoperative radiotherapy.
* Signed informed consent

Exclusion Criteria:

* the patients whose preoperative evaluation is below T3 stage with middle and rectal cancer.
* Active internal bleeding (such as gastrointestinal bleeding), urogenital system, or have not cure of peptic ulcer in four weeks
* Severe liver and kidney dysfunction
* Intracranial tumor, suspicious aortic dissection, arteriovenous malformation, aneurysm
* Thrombolysis treatment in one week
* Allergies of thrombolysis drug or contrast
* Participated in any clinical trials within three months

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-01-01 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Decide and record the region of radiotherapy | Intraoperation
  The operator will confirm and record the range of intrabeam after removal of tumor such as the length and height to modify the dose and the time of intrabeam.
The basic information and medical history achieved (questionnaire) | baseline
  Investigators will take a overall information about the patients including the physical condition,history of present illness,family genetic history etc;Then the information will be recorded in a format to develop a statistic analysis.

SECONDARY OUTCOMES:
Major Adverse Events | 1 year after operation
  The local relapse (pelvic pain, bleeding and intestinal obstruction included)or metastasis will be recorded by the investigator
The short-term complications | 1 year after operation
  The short-term complications(seroma,wound dehiscence and bleeding hematomas)will be followed up by investigator.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: Yes
When the investigators complete the study and publish our data.
Supporting Information: Study Protocol, CSR
Time Frame: When the investigators complete the study and publish our data.